CLINICAL TRIAL: NCT01413373
Title: Clinical Validation of the Three-dimensional Computer Tomography Based Craniofacial Cephalometric Analysis
Brief Title: 3D Craniofacial Cephalometric Analysis
Acronym: ACRO3D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: B40320083938; 2014/13MAR/104 (Other: CEHF); MAXILLARY SEPTA 3D (Other: CLAIRE)
Record Dates: First submitted 2011-07-20; First posted 2011-08-10 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Malocclusion
Keywords: cephalometry; three-dimensional; CT scan; lateral radiography; facial symmetry; maxillomandibular dysmorphoses
MeSH Terms: conditions — Malocclusion | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: cone beam computed tomography — A preoperative CBCT is performed for all patients in this study for medical reason
  Other Names: medical imaging, CBCT
Radiation: computer tomography — One cone beam computer tomography examination before surgery
  Other Names: medical imaging

SUMMARY:
Development of three-dimensional craniofacial cephalometric analysis for virtual planning in orthognathic surgery.

DETAILED DESCRIPTION:
Cone beam computed tomography is taken for diagnosis independently from this study. Investigators are using this medical imaging for performing the 3D cephalometric analysis. Investigators apply a set of well described landmarks of three-dimensional reconstruction of the skull from patients suffering from diverse craniofacial malformations. Then a set of specific measurements is taken from the patient and provide insights how to modify the anatomy of the patient to improve the skull's architecture and symmetry

ELIGIBILITY:
Inclusion Criteria:

* maxillomandibular dysmorphoses,
* facial asymmetry,
* craniofacial syndromes

Exclusion Criteria:

* patients with orthodontic treatment only
* growing patients

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient more than 18 yeras old, no pregnant women, no child
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2008-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
topological description of maxillomandibular dysmorphosis (angles, distances) | 2014
  Anterior cranial base angle on three-dimensional CT recostruction of the skull (in degrees) Posterior cranial base angle on three-dimensional CT recostruction of the skull (in degrees) Ratio between distance from nasion to anterior nasal spine/anterior nasal spine to chin landmark (without unit of maesurment) Measurements between various anatomic landmarks for orbits and maxillary sinus structures on the three-dimensional CT reconstruction of the patient's skull (in mm).

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Olszewski, DDS,MD,PhD, Principal Investigator — Department of Oral and maxillofacial surgery, Cliniques Universitaires saint Luc
Locations (1):
- Department of oral and maxillofacial surgery, Cliniques universitaires saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No